CLINICAL TRIAL: NCT02141217
Title: Efficacy, Safety and Tolerability of Amoxicillin + Clavulanic Acid (875mg/125mg) Two Times a Day Compared to Clindamycin (150mg) Four Times a Day for 5-7 Days in Treatment of Acute Odontogenic Infection With or Without Abscess
Brief Title: AUGMENTIN™ in Dental Infections
Acronym: AUGDENT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 117044
Record Dates: First submitted 2014-05-15; First posted 2014-05-19 (Estimated); Results first posted 2014-08-28 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-08

CONDITIONS: Focal Infection, Dental
Keywords: Odontogenic (Dental) Infections; Dental infections, periapical abscess; Bacterial infection
MeSH Terms: conditions — Focal Infection, Dental; Infections; Periapical Abscess; Bacterial Infections | interventions — Amoxicillin-Potassium Clavulanate Combination; Clindamycin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Amoxicillin/clavulanate (Active Comparator): Amoxicillin/ clavulanate 1 g bd for for at least 5 days upto seven days depending on treament response
  Interventions: Drug: Amoxicillin/clavulanate
- Clindamycin (Active Comparator): Clindamycin 150 mg qid for at least 5 days or maximum 7 days depending upon treatment response
  Interventions: Drug: Clindamycin

INTERVENTIONS:
Drug: Amoxicillin/clavulanate — Amoxicillin/clavulanate 1 g bd for at least 5 days or maximum 7 days depending upon the treatment response.
  Arms: Amoxicillin/clavulanate
Drug: Clindamycin — Clindamycin 150 mg qid for at least 5 days or maximum 7 days depending upon the treatment response.
  Arms: Clindamycin

SUMMARY:
In clinical practice, amoxicillin + clavulanic acid is widely used in the treatment of odontogenic infection. Therefore, this study is designed to generate data to support its use by demonstrating efficacy, safety and tolerability in comparison with clindamycin in subjects with acute odontogenic infections with or without abscess. This will be a two-arm, parallel, comparative, observer blind, randomised study to assess efficacy, safety and tolerability of amoxicillin + clavulanic acid (875mg/125mg) in comparison with clindamycin (150mg) administered for 5-7 days in subjects with acute odontogenic infections with or without abscess. The study will be performed in adult subjects both male and female ≥18 years of age who present with acute odontogenic infections. A total of 472 subjects will be randomized in 1:1 ratio, i.e. 236 subjects in each treatment arm. The treatment duration of the study will be at least 5 days or maximum 7 days depending upon the treatment response. Subjects will be assessed on Day 5 and if Investigator feels the need of continuing the treatment at Day 5 then treatment will be continued till Day 7. For subjects who do not show treatment response on Day 5, assessments will be performed on Day 7.

DETAILED DESCRIPTION:
This two-arm, parallel, comparative, observer blind, randomised study will be performed in adult subjects both male and female ≥18 years of age who present with acute odontogenic infection with or without abscess. A total of 472 subjects will be randomised in 1:1 ratio to get 205 evaluable subjects in each study arm. After obtaining informed consent, subject will undergo surgical intervention including surgical incisions, drainages, removal of the involved tooth, debridement, puncture lavage or trephination, if deemed necessary by the Investigator. These surgical interventions will be performed before the start of study treatment. On Day 0 after confirming the eligibility, subjects will be randomised to either of the study arms. The treatment duration of the study will be at least 5 days which may increase to 7 days, if Investigator feels the need of continuing the treatment at Day 5. In such cases clinical assessment will be done again at Day 7. Thus the efficacy evaluation will be performed at baseline (Day 0) prior to study drug administration and on Day 5 and/ or 7. Safety laboratory evaluations will be performed at Screening Visit and will be repeated at end of study treatment i.e. either on Day 5 or Day 7. On Baseline, Day 2, Day 5 and/ or Day 7, Visual Analogue Scale (VAS) will be used to measure amount of pain and swelling that a subject will experience. This scale has numerical ratings from 0 to 10. Zero would mean "No pain" and 10 would mean "Worst possible pain". The subject will be asked to choose the most appropriate score on VAS which best describes his/her pain status over last 24 hours. While using VAS for swelling, zero would mean "No swelling" and 10 would mean "Maximum possible swelling". The Investigator will choose the most appropriate score on VAS which best describes subject's swelling.

Sample for microbiological culture will be obtained at the discretion of Investigator while performing the surgical procedure. When microbiological culture is indicated and feasible, two sets (each consisting of aerobic and anaerobic media) will be obtained. This sampling will be done in approximately 80 subjects randomly who will provide consent at Screening. The sample will be collected and dispatched in appropriate transport medium to the central laboratory for culture and antibiotic susceptibility.

Protocol waivers or exemptions will not be allowed.

The total duration of each subject's participation will be 6-9 days including Screening period of 0-1 day (Day -1 to Day 0) and Treatment period of 5-7 days (Day 0 to Day 5-7).

The primary objective of the study is to compare clinical efficacy (cure and improvement) of both the treatment arms which uses VAS for assessment of pain and swelling. Since the clinical efficacy parameters are subjective, it is mandatory to keep the observer/Investigator blinded during the study assessment. In addition, designing blinded study is challenging owing to different dosage regimen and formulation of study drugs. The study design of double blind double dummy is not recommended in view of increased pill burden which in turn can have an impact on treatment compliance. The possibility of over-encapsulation is ruled out due to large pill size of amoxicillin + clavulanic acid. Therefore to maintain blinding of Investigators, the study is designed as observer blind with Investigator remaining blinded throughout the study period. An unblinded study team member will be appointed for each site who will be involved in dispensing of the study drugs to subjects. The unblinded study team member will remain present during subject assessment for all study visits and will ensure that Investigator remains blinded to treatment assignment.

Study treatment includes amoxicillin + clavulanic acid (875mg/125mg) two times daily or clindamycin (150mg) four times daily for 5-7 days both administered orally with meal. Augmentin™ (amoxicillin + clavulanic acid) from GSK and Dalacin-C (clindamycin) from Pfizer will be used as study treatments. The contents of the label will be in accordance with all applicable regulatory requirements.

Patients can receive additional medical therapy such as analgesics or anti-inflammatory drugs. However, opioid analgesics and any other antibiotic apart from study drugs will not be permitted during entire study period.

This study will be conducted in accordance with ICH GCP, all applicable subject privacy requirements, and the ethical principles that are outlined in the Declaration of Helsinki 2008, including IRB/ IEC review and approval of study protocol and any subsequent amendments, subject informed consent and Investigator reporting requirements.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criterion:

  * Adult (≥18 years of age) males and females
  * Subjects with diagnosis of acute odontogenic infections of following types requiring antibiotic therapy
* Periapical abscess
* Aute periodontitis
* Pericoronitis • Provision of voluntary written informed consent

Exclusion Criteria:

* Subjects presenting with complications like osteomyelitis, dentocutaneous fistula, dentoalveolar fistula, draining sinus, facial-space swelling, necrotizing fasciitis OR subjects requiring hospitalization, aggressive intravenous antimicrobial therapy, requiring local application of antimicrobials for the treatment of odontogenic infection.
* Subjects presenting with odontogenic infections secondary to traumatic injury to the face.
* Subjects with valvular heart disease, prosthetic heart valves, congenital heart disease or any other conditions prone to infective endocarditis
* Subjects with a known clinically significant abnormality identified at screening on physical examination or known laboratory tests which, in the judgment of the Investigator, would preclude safe completion of the study
* Subject who has taken a systemic antibiotic within 2 weeks before study drug administration or a long-acting injectable antibiotic (e.g., penicillin G benzathine) within 4 weeks before study drug administration
* Immunocompromised subjects or subjects on immunosuppressants or systemic corticosteroids
* Subjects with chronic gingivitis or chronic periodontitis
* Subjects with uncontrolled diabetes mellitus or HIV infection
* History of hypersensitivity or allergic reactions to any beta-lactam such as penicillin, cephalosporin, moxicillin/clavulanic acid or clindamycin
* Concomitant infection, that requires additional antimicrobial therapy during the study period
* Subjects with clinically significant liver disease as defined by alanine aminotransferase (ALT) or aspartate minotransferase (AST) levels >2.5 times the upper limit of normal (ULN) or a diagnosis of chronic active hepatitis including that of viral etiology, or on antiviral or immunosuppressive therapy.
* Subjects with renal impairment with serum creatinine > 1.7 mg/dl in men and >1.5mg/dl in women.
* Subjects with infectious mononucleosis
* Subjects with history of documented Clostridium difficile-associated diarrhoea or existing diarrhoea
* Concomitant treatment with oral anticoagulants, methotrexate or probenicid
* Female subjects of childbearing potential in whom pregnancy cannot be excluded by a negative pregnancy test and who are not using reliable method of contraception
* Subjects with lactose intolerance or Lapp lactase deficiency or glucose-galactose malabsorption
* Pregnant or lactating female subjects

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 472 (Actual)
Dates: Start 2013-03-21 (Actual); Primary Completion 2013-12-28 (Actual); Study Completion 2013-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (12):
- Malaysia (4):
  - GSK Investigational Site, Kuala Lumpur
  - GSK Investigational Site, Kuala Selangor
  - GSK Investigational Site, Perak
  - GSK Investigational Site, Putrajaya
- Philippines (3):
  - GSK Investigational Site, Cebu
  - GSK Investigational Site, Davao City
  - GSK Investigational Site, Quezon
- Thailand (3):
  - GSK Investigational Site, Lampang
  - GSK Investigational Site, Pran Buri
  - GSK Investigational Site, Songkhla
- Vietnam (2):
  - GSK Investigational Site, Hanoi
  - GSK Investigational Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Tancawan AL, Pato MN, Abidin KZ, Asari AS, Thong TX, Kochhar P, Muganurmath C, Twynholm M, Barker K. Amoxicillin/Clavulanic Acid for the Treatment of Odontogenic Infections: A Randomised Study Comparing Efficacy and Tolerability versus Clindamycin. Int J Dent. 2015;2015:472470. doi: 10.1155/2015/472470. Epub 2015 Aug 2. PMID 26300919
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 117044 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 117044 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 117044 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 117044 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 117044 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 117044 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 510 participants (par.) were screened; 472 were randomized to receive one of the two study treatments. Of the 472 par.; 235 par. were randomized to the amoxicillin + clavulanic acid (amx+clv) arm and 237 par. to the clindamycin (clin) arm.
Pre-assignment Details: Amongst the randomized par., 236 par. received amx+clv and 235 par. received clin as 2 par. randomized to the clin arm incorrectly received amx+clv and 1 par. randomized to amx+clv arm confirmed not consuming even a single dose of study drug.
Groups:
- Amoxicillin 875 mg + Clavulanic Acid 125 mg: Participants received amoxicillin 875 milligrams (mg) plus clavulanic acid 125 mg orally twice daily with meals for a duration of five to seven days in participants with acute odontogenic infection with or without abscess.
- Clindamycin 150 mg: Participants received clindamycin 150 mg orally four times daily for a duration of five to seven days in participants with acute odontogenic infection with or without abscess.
Period: Overall Study
Arm/Group | Amoxicillin 875 mg + Clavulanic Acid 125 mg | Clindamycin 150 mg
Started | 234 | 237
ITT Population-Randomized Treatment Arm | 234 | 237
ITT Population-Actual Treatment Received | 236 | 235
Completed | 223 | 229
Not Completed | 11 | 8
Not completed — Adverse Event | 1 | 2
Not completed — Protocol Violation | 1 | 4
Not completed — Withdrawal by Subject | 6 | 0
Not completed — Lost to Follow-up | 1 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Surgical Intervention | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Amoxicillin 875 mg + Clavulanic Acid 125 mg: Participants received amoxicillin 875 mg plus clavulanic acid 125 mg orally twice daily with meals for a duration of five to seven days in participants with acute odontogenic infection with or without abscess.
- Total: Total of all reporting groups
Arm/Group | Amoxicillin 875 mg + Clavulanic Acid 125 mg | Clindamycin 150 mg | Total
Number analyzed (Participants) | 234 | 237 | 471
Age, Continuous [Mean (Standard Deviation); unit: Years] — Amongst the randomized par., 236 par. received amx+clv and 235 par. received clin as 2 par. randomized to the clin arm incorrectly received amx+clv and 1 par. randomized to amx+clv arm confirmed not consuming even a single dose of study drug.
  Years | 33.1 (12.8) | 32.6 (12.0) | 32.9 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Amongst the randomized par., 236 par. received amx+clv and 235 par. received clin as 2 par. randomized to the clin arm incorrectly received amx+clv and 1 par. randomized to amx+clv arm confirmed not consuming even a single dose of study drug.
  Participants
    Female | 135 | 143 | 278
    Male | 99 | 94 | 193
Race/Ethnicity, Customized [Number; unit: Participants] — Amongst the randomized par., 236 par. received amx+clv and 235 par. received clin as 2 par. randomized to the clin arm incorrectly received amx+clv and 1 par. randomized to amx+clv arm confirmed not consuming even a single dose of study drug.
  Participants
    Asian-Central/South Asian Heritage | 0 | 1 | 1
    Asian-East Asian Heritage | 1 | 4 | 5
    Asian-South East Asian Heritage | 233 | 232 | 465

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Clinical Success (Cure or Improvement) Considering Clinical Judgment of the Investigator at the End of Treatment (Day 5 or Day 7)
Description: Clinical success is defined as the achievement of cure or improvement in signs and symptoms of odontogenic infections. Cure is defined as the complete resolution of signs and symptoms of infection present at baseline, such that no additional antimicrobial therapy is required. Improvement is defined as the resolution of fever (if present at baseline), >70% reduction in swelling and pain and improvement in other signs and symptoms such that no additional antimicrobial therapy is required. Visual Analogue Scale (VAS) is used to measure the amount of pain and swelling that a participant experiences. This scale has numerical ratings from 0 to 10. Zero indicates no pain and 10 indicates worst possible pain.
Time Frame: Day 5 or Day 7 [End of treatment]
Population: Per-Protocol (PP) Population: all participants in the Intent-to-Treat (ITT) Population (defined as all randomized participants who received at least one dose of study medication) who were without major protocol violations and had end of treatment clinical response assessment available.
Measure: Number; unit: Percentage of participants
Arm/Group | Amoxicillin 875 mg + Clavulanic Acid 125 mg | Clindamycin 150 mg
Number analyzed (Participants) | 211 | 203
Percentage of participants | 88.2 | 89.7
Statistical Analysis 1: Comparison: Amoxicillin 875 mg + Clavulanic Acid 125 mg vs Clindamycin 150 mg; Test type: Non-Inferiority or Equivalence — The assessment of non-inferiority was based on Farrington and Manning method. The upper limit of two-sided 95% confidence interval of less than 10 % provide enough evidence to show the non-inferiority between the treatment arms; Treatment Difference (percentage) = 1.5, 95% CI 2-sided [-4.9 to 8.0]

2. Primary Outcome: Percentage of Participants Achieving Clinical Success (Cure or Improvement) Considering Clinical Judgment of the Investigator at the End of Treatment (Day 5 or Day 7)
Description: as for outcome 1
Time Frame: Day 5 or Day 7 [End of treatment]
Population: Intent-To-Treat-Efficacy (ITT-E) Population: all participants in the ITT participants who had at least one post-Baseline assessment of clinical success response (clinical response based on assessment on odontogenic infection and VAS Score).
Measure: Number; unit: Percentage of participants
Arm/Group | Amoxicillin 875 mg + Clavulanic Acid 125 mg | Clindamycin 150 mg
Number analyzed (Participants) | 228 | 235
Percentage of participants | 85.5 | 86.4
Statistical Analysis 1: Comparison: Amoxicillin 875 mg + Clavulanic Acid 125 mg vs Clindamycin 150 mg; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Treatment Difference (percentage) = 0.9, 95% CI 2-sided [-5.6 to 7.4]

3. Primary Outcome: Percentage of Participants Achieving Clinical Success (Cure or Improvement) Considering Clinical Judgment of the Investigator at the End of Treatment (Day 5 or Day 7)
Description: as for outcome 1
Time Frame: Day 5 or Day 7 [End of treatment]
Population: Intent-to-Treat (ITT) Population (randomized as per treatment allocation): all randomized participants who received at least one dose of study medication. If the post-Baseline assessment of clinical success response was missing then "Clinical Success" is considered as "No" i.e. the participant was treated as "Clinical Failure".
Measure: Number; unit: Percentage of participants
Groups:
- Amoxicillin 875 mg + Clavulanic Acid 125 mg: Participants randomized to amoxicillin 875 mg plus clavulanic acid 125 mg.
- Clindamycin 150 mg: Participants randomized to clindamycin 150 mg.
Arm/Group | Amoxicillin 875 mg + Clavulanic Acid 125 mg | Clindamycin 150 mg
Number analyzed (Participants) | 234 | 237
Percentage of participants | 83.3 | 85.7
Statistical Analysis 1: Comparison: Amoxicillin 875 mg + Clavulanic Acid 125 mg vs Clindamycin 150 mg; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Treatment Difference (percentage) = 2.3, 95% CI 2-sided [-4.4 to 9.0]

4. Secondary Outcome: Number of Participants Achieving Clinical Success (Cure or Improvement) Considering Clinical Judgment of the Investigator at Day 5
Description: as for outcome 1
Time Frame: Day 5
Population: ITT-E Population. Only the participants with Day 5 assessments were considered for analysis.
Measure: Number; unit: Participants
Arm/Group | Amoxicillin 875 mg + Clavulanic Acid 125 mg | Clindamycin 150 mg
Number analyzed (Participants) | 220 | 230
Participants | 169 | 159

5. Secondary Outcome: Number of Participants (Par.) Achieving Clinical Success (CS) (Cure or Improvement [Imp] in Signs [s] and Symptoms [sx] [s/sx]) Without Considering Clinical (cl) Judgment (Jdg) of the Investigator (Inv) at Day 5
Description: CS is defined as cure or imp in s/sx of odontogenic infections. Cure is defined as the complete resolution of s/sx of infection present at Baseline (BL) and imp is defined as resolution of fever (if present at BL), >70% reduction in swelling and pain and imp in other s/sx such that no additional antimicrobial (ant) therapy is required. In event of cure or imp with complete resolution of fever and >70% reduction in swelling and pain, but 'no change' or 'worsening from BL' in other s/sx (like increased leucocyte count/tooth mobility), the inv's opinion was sought on whether additional ant therapy was required. Par. that required no additional ant therapy were considered a 'success' while those requiring additional ant therapy were deemed a 'failure'. For a sensitivity analysis, all such par. with 'no change' or 'worsening from BL' in these other s/sx were considered as cl failures and termed 'Without Considering Cl Jdg of Inv', even though main s/sx are 'cured' or 'improved'. .
Time Frame: Day 5
Population: ITT-E Population
Measure: Number; unit: Participants
Arm/Group | Amoxicillin 875 mg + Clavulanic Acid 125 mg | Clindamycin 150 mg
Number analyzed (Participants) | 220 | 230
Participants | 158 | 150

6. Secondary Outcome: Change From Baseline in the Visual Analogue Scale Assessment of Pain Score at Days 2, 5 and 7
Description: Visual Analogue Scale (VAS) is used to measure the amount of pain that the participant experiences. This scale has numerical ratings from 0 to 10. Zero indicates no pain and 10 indicates worst possible pain. Change in Pain/Swelling is calculated as VAS score at Baseline minus the score at a later time point (Day 2, 5 or 7).
Time Frame: Baseline, Days 2, 5 and 7
Population: ITT-E Population. Only those participants available indicated time points were analyzed (represented by n=X, X in the category titles). Different participants may have been analyzed at different time points, so the overall number of participants analyzed reflects everyone in the ITT-E population.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Amoxicillin 875 mg + Clavulanic Acid 125 mg | Clindamycin 150 mg
Number analyzed (Participants) | 228 | 235
Scores on a scale
  Day 2, n=227, 233 | 3.34 [3.08 to 3.61] | 3.07 [2.81 to 3.33]
  Day 5, n=219, 228 | 5.49 [5.27 to 5.71] | 5.38 [5.16 to 5.60]
  Day 7, n=57, 71 | 6.38 [6.02 to 6.74] | 6.34 [6.02 to 6.66]

7. Secondary Outcome: Change From Baseline in Visual Analogue Scale Assessment of Swelling at Days 2, 5 and 7
Description: Visual Analogue Scale (VAS) is used to measure the amount of swelling that the participant experiences. This scale has numerical ratings from 0 to 10. Zero indicates no swelling and 10 indicates worst possible swelling. Change in Pain/Swelling is calculated as VAS score at Baseline minus the score at a later time point (Day 2, 5 or 7).
Time Frame: Baseline, Days 2, 5 and 7
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Amoxicillin 875 mg + Clavulanic Acid 125 mg | Clindamycin 150 mg
Number analyzed (Participants) | 228 | 235
Scores on a scale
  Day 2, n=219, 225 | 1.92 [1.72 to 2.11] | 1.61 [1.42 to 1.80]
  Day 5, n=214, 223 | 3.68 [3.51 to 3.85] | 3.60 [3.43 to 3.76]
  Day 7, n=55, 68 | 4.21 [3.94 to 4.49] | 4.61 [4.36 to 4.86]

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the Baseline (Day 0) until the last dose of study drug (Day 7) or early withdrawal (average of Day 5.88).
Description: SAEs and non-serious AEs were collected in members of the ITT Population, comprised of all randomized participants who received at least one dose of investigational product , according to the actual treatment received.
Arm/Group | Amoxicillin 875 mg + Clavulanic Acid 125 mg | Clindamycin 150 mg
Serious Adverse Events (participants affected / at risk) | 0/236 | 0/235
Other Adverse Events (participants affected / at risk) | 99/236 | 93/235
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Amoxicillin 875 mg + Clavulanic Acid 125 mg (N=236) | Clindamycin 150 mg (N=235)
Abdominal discomfort (Gastrointestinal disorders) | 11 | 7
Diarrhoea (Gastrointestinal disorders) | 19 | 28
Alanine aminotransferase increased (Investigations) | 26 | 24
Aspartate aminotransferase decreased (Investigations) | 8 | 2
Aspartate aminotransferase increased (Investigations) | 24 | 20
Blood bilirubin increased (Investigations) | 12 | 13
Increased appetite (Metabolism and nutrition disorders) | 20 | 15
Dizziness (Nervous system disorders) | 18 | 14
Headache (Nervous system disorders) | 8 | 14
Somnolence (Nervous system disorders) | 19 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.